CLINICAL TRIAL: NCT01947127
Title: Can Venous Lactate Predict the Progression to Overt Septic Shock and Mortality in Non-elderly Sepsis Patients Without Hemodynamic Shock in Emergency Department?
Brief Title: Venous Lactate in Progression to Overt Septic Shock and Mortality in Non-elderly Sepsis Patients in Emergency Department
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Khrongwong Musikatavorn, MD., Khrongwong Musikatavorn, MD, Chulalongkorn University
Other Study IDs: 793/2012
Record Dates: First submitted 2013-09-10; First posted 2013-09-20 (Estimated); Results first posted 2015-05-07 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2015-04

CONDITIONS: Sepsis; Disease Progression; Septic Shock; Fatal Outcome
Keywords: Lactate; Sepsis; Septic shock; Disease progression; Prognosis
MeSH Terms: conditions — Sepsis; Disease Progression; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Venous blood lactate obtained by standard venipuncture together with other essential blood works before giving antibiotics or intravenous fluid, if required. Lactate level is measured by Epoc® point-of-care blood analyzer (Epocal Inc., Ottawa, ON, Canada) within 5 minutes after obtaining the venous sample without any preservative.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- High lactate: Initial venous lactate level equal to or more than 2.0 mmol/L
- Low lactate: Initial venous lactate level less than 2.0 mmol/L

SUMMARY:
To investigate the role of initial venous lactate in predicting the severity progression to overt septic shock and 30-day mortality in non-elderly patients without hemodynamic shock who suspected to have acute infections.

DETAILED DESCRIPTION:
Blood lactate is one of the markers that can predict the organ failures and mortality in emergency department (ED) patients with sepsis. Regarding its predictive role in the clinical deterioration in normotensive sepsis patients, a recent prospective observational study of the patients with moderately-high serum lactate (2.0-3.9 mmol/L) showed that one-forth of the patients eventually developed progressive organ dysfunctions or required vasopressor or mechanical ventilator. Unfortunately, low serum lactate (< 2.5 mmol/L) was still found up to 50% of overt septic shock patients, even in vasopressor-dependent cases. For the prognostic role on mortality, numbers of articles showed that blood lactate can also predict death in sepsis patients, especially in those who are elderly and critically-ill. However, no previous study was done in younger patients since lactate kinetics in the body may differ among the age groups. The primary aim of our study is to investigate the role of initial venous lactate levels in predicting the chance of severity progression to overt septic shock especially in non-elderly patients who suspected to have acute infections and without hemodynamic shock in ED. The secondary outcomes are to evaluate its prognostic role on hospital length of stay and 30-day mortality of this target population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Confirmed or suspected diagnoses of acute infections (within 7 days)
* Major infections (e.g. Acute pyelonephritis, Acute bronchitis/pneumonia, Acute hepatobiliary tract infections, intrabdominal abscesses, meningitis and other central nervous system infections, soft tissue infections involving more than 10 square centimeters of the skin surface or deeper down beyond the dermis, significant tropical infections; dengue fever, leptospirosis, typhus fevers, or high fever from any infectious sources)
* Systolic blood pressure more than 90 mmHg at presentation
* Mean arterial pressure more than 70 mmHg at presentation

Exclusion Criteria:

* Duplicated cases that have participated in this study during the study period
* Overt organ hypoperfusion (e.g. cold, clammy or mottling skin, altered mental status; Glasgow Coma Scale equal to or less than 12 or decrease > 1 compared with the baseline)
* Pulse oximetry equal to or less than 90% at ambient air
* received intravenous fluid more than 10 ml/kg prior to the venous blood sampling
* received intravenous antibiotics for more than 1 hours prior to the venous blood sampling
* Minor infections (e.g. uncomplicated upper respiratory tract infections, gastroenteritis, minor skin infections)
* currently taking antiretroviral drugs
* having or suspicious of having seizures in the past 72 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patients of King Chulalongkorn Memorial Hospital (a 1500-bed, tertiary-care, university-affiliated urban hospital)
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khrongwong Musikatavorn, MD, Principal Investigator — Department of Medicine, Facalty of medicine, Chulalongkorn University
Locations (1):
- Emergency Medicine Unit, King Chulalongkorn Memorial Hospital, Patumwan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Musikatavorn K, Thepnimitra S, Komindr A, Puttaphaisan P, Rojanasarntikul D. Venous lactate in predicting the need for intensive care unit and mortality among nonelderly sepsis patients with stable hemodynamic. Am J Emerg Med. 2015 Jul;33(7):925-30. doi: 10.1016/j.ajem.2015.04.010. Epub 2015 Apr 10. PMID 25936479

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started at April 2013 to October 2014 at King Chulalongkorn Memorial Hospital, a university-affiliated, 1,500 bed, tertiary care urban hospital
Period: Overall Study
Arm/Group | High Lactate | Low Lactate
Started | 166 | 292
Completed | 143 | 249
Not Completed | 23 | 43
Not completed — Protocol Violation | 18 | 38
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Data loss | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Lactate | Low Lactate | Total
Number analyzed (Participants) | 143 | 249 | 392
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 143 | 249 | 392
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (13.7) | 42.8 (14.4) | 44.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 120 | 184
  Male | 79 | 129 | 208
Race/Ethnicity, Customized [Number; unit: participants]
  Thai and Southeast Asian | 143 | 249 | 392
Region of Enrollment [Number; unit: participants]
  Thailand | 143 | 249 | 392

OUTCOME MEASURES:

1. Primary Outcome: Proportion of the Patients Who Require Vasopressor/Mechanical Ventilator
Description: Proportion of the patients in each cohort who require vasopressor/mechanical ventilator to maintain their vital signs in the next 72 hours after venous lactate measurement.
Time Frame: 72 hours after venous lactate measurement
Measure: Number; unit: participants
Arm/Group | High Lactate | Low Lactate
Number analyzed (Participants) | 143 | 249
participants | 53 | 21

2. Secondary Outcome: All-cause Mortality Rates
Description: Electronic database retrieval of in- and outpatient clinical records together with telephone follow-ups to the patients or their contact personnel are employed to every case in the next 30 days after the day of presentation to the emergency department to identify the deceased cases. All-cause mortality rates of each cohort will be compared by the survival analysis.
Time Frame: 30 days after the day of presentation to the emergency department
Population: Four patients out of 392 patients were excluded from secondary (mortality) outcome analysis due to unknown mortality status. As a result, 388 patients (139 in high lactate group and 249 in low lactate group) were available for mortality outcome analysis.
Measure: Number; unit: participants
Arm/Group | High Lactate | Low Lactate
Number analyzed (Participants) | 139 | 249
participants | 18 | 13

3. Secondary Outcome: Hospital Length of Stay
Description: Numbers of days spent in the hospital since the emergency department arrival to hospital discharge
Time Frame: Patients will be followed for the duration of hospital stay, an expected average of 7 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | High Lactate | Low Lactate
Number analyzed (Participants) | 143 | 249
Days | 6 [2 to 14] | 3 [2 to 8]

ADVERSE EVENTS:
Time Frame: Overall study period
Arm/Group | High Lactate | Low Lactate
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/249
Other Adverse Events (participants affected / at risk) | 0/143 | 0/249

LIMITATIONS AND CAVEATS:
1. This was an observational study that did not evaluate the aggressiveness of the treatment strategies. 2. The study was done in a single, urban, university hospital. 3. The staging of co-morbidity (e.g. cancers) was not well-categorized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes